CLINICAL TRIAL: NCT06420362
Title: Examination of the Effect of Exercise Training With Upper Extremity Blood Flow Restriction on Upper Extremity Muscle Strength and Performance in Basketball Players
Brief Title: Blood Flow Restriction Training in Basketball Players
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Buket AKINCI, Assoc.Prof., Biruni University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 80-23-05
Record Dates: First submitted 2024-05-09; First posted 2024-05-20 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Basketball Players
Keywords: bloodflowrestriction; basketball; basketball performance; kaatsu training
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood Flow Restriction Training Group (Experimental): While the basketball players continue their current basketball training; The 90-minute BFR program will be applied 3 sessions a week for 3 weeks. In the BFR program, biceps curls, triceps curls, shoulder presses, shoulder abduction exercises and sport-specific routine training will be applied. Exercises: 30% of 1 maximum repetition with resistance and 60% of arterial occlusion pressure restricted; Based on previous studies in the literature, the first set will be performed with 30 repetitions and the other three sets with 15 repetitions, a total of 4 sets and a 30-second rest between sets. There will be a 10-minute warm-up exercise before each BFR training and a 10-minute cool-down exercise at the end of the training.
  Interventions: Other: Blood Flow Restriction
- Routine Training (No Intervention): Initial evaluations will be made for all participants. Then, they will continue their routine basketball training programs for 3 weeks.

INTERVENTIONS:
Other: Blood Flow Restriction — Before BFR training, a repetition maximal (1-RM) test will be determined by selecting a weight with which athletes can perform a maximum of 10 repetitions. The number of repetitions obtained here and the weight lifted will be written into the Brzycki formula, whose validity and reliability has been proven, and 1-TM will be calculated.
  Brzycki formula; 1-TM = [100 x (Weight Lifted) / [(102.78 - 2.78 x (Number of Reps)] The arterial occlusion pressure of the participants will be measured with a Doppler Ultrasound device by increasing the cuff to the point where the auscultatory pulse of the brachial artery ceases until occlusion occurs in the brachial artery. Then, 60% of this value will be calculated and BFR will be performed during the exercises.
  Arms: Blood Flow Restriction Training Group

SUMMARY:
Blood Flow Restrictive Exercises (BFR) provide strength increase with less load than required for traditional muscle strengthening and power. As an alternative for populations that have difficulty training with high loads and speeds, low-intensity BFR training has been shown to improve muscle strength and aerobic parameters and to be safe, even in professional athletes and individuals with chronic diseases in various populations. The aim of our study is to examine the effects of BFR applied to the upper extremity on upper extremity muscle strength and performance in basketball players.

DETAILED DESCRIPTION:
Basketball is a demanding sport that requires participants to display a high level of physical fitness and special sporting skills. Basketball requires a high level of anaerobic and aerobic conditioning and is not only a team sport, but also a sport that requires players to demonstrate their individual characteristics. In this regard, it is thought that the determination of performance components based on field tests is a more suitable method for determining the athletic levels of athletes with special needs.

BFR, which aims to restrict blood flow to the muscle during exercise, is traditionally known as 'kaatsu'. Blood flow is restricted with a pressure-controlled and monitorable exercise belt produced for BFR. In order for the method to be successful, the tourniquet method must be applied to the proximal region of the extremity, and in this way, less blood flow to the muscle can actually be achieved.

With BFR, it is recommended that the external pressure be made sufficient to restrict the arterial oxygen pressure between 40% and 80%, and it is thought that the effects of exercise increase in this hypoxic environment. In this way, it is sufficient to perform the exercises at 20% to 40% of the 1 maximum repetition, not 60-85%, which is normally required for muscle hypertrophy. An ischemic and hypoxic muscle environment during BFR; It has been hypothesized that it is produced to cause high levels of metabolic stress and mechanical tension. Both metabolic stress and mechanical tension have been described as "primary hypertrophy factors" and are theorized to activate other mechanisms for muscle growth.

Strength training performed by restricting blood flow plays an important role in muscle hypertrophy by activating the endocrine system. It has been proven that low-intensity blood flow restriction training increases the plasma concentration of growth hormone more than normal exercises. BFR involves low-intensity resistance training and is placed on the proximal portion of the lower or upper extremity muscles to be worked with a bandage or cuff that restricts blood flow, providing appropriate superficial pressure.

The aim of this study is to examine the effects of BFR applied to the upper extremity on upper extremity muscle strength and performance in basketball players.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-25,
* Having been attending training regularly for at least one year,
* Having been playing basketball as a licensed player for at least 3 months,
* Male athletes,
* Volunteering to participate in the study

Exclusion Criteria:

* Individuals with orthopedic or neurological disabilities that may prevent the exercise test,
* Individuals who have had a sports injury in the last 6 months,
* Not actively participating in training,
* Taking a break from sports
* Individuals with inadequate cooperation

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Bench press test | Change from Baseline Bench press test at 3 weeks and 6 weeks
  Bench Press 1RM test will be applied for upper extremity muscle strength. the athlete's 1RM weight will be determined.
Hand Grip Strength | Change from Baseline Hand Grip Strength at 3 weeks and 6 weeks
  "Jamar (NY 10533)" brand dynamometer, one of the hydraulic measuring instruments, will be used to measure grip force.

SECONDARY OUTCOMES:
20 m Sprint Test | Change from Baseline Bench press test at 3 weeks and 6 weeks
  A 20 m speed test will be applied to evaluate the speed of the participants. Running basketball players will be asked to run the 20-meter track at maximum level after starting.
T Agility Test | Change from Baseline T Agility Test at 3 weeks and 6 weeks
  T test will be applied to evaluate the agility of the participants.The best time of the participants will be recorded.
Free Throw Test | Change from Baseline Free Throw Test at 3 weeks and 6 weeks
  A shooting test will be applied to evaluate the shooting skills of the athletes. Athletes will be asked to make 2 sets of free throws with 8 repetitions after the "Start" command from the starting position behind the foul (free throw) line. Total scores will be recorded at the end of the test.
Fatigue Assessment | immediately after each BFR session
  The modified Borg CR10 scale will be used to evaluate perceived fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Buket AKINCI, Assoc.Prof., Study Chair — Biruni University
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The data will be shared during the publication process if the journal will ask.